CLINICAL TRIAL: NCT04540900
Title: A Phase I Study of KB301, a Replication-Incompetent, Non-Integrating Vector Expressing Human Type III Collagen (COL3) for the Treatment of Superficial Skin Depressions
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Krystal Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEARL-1
Record Dates: First submitted 2020-08-19; First posted 2020-09-07 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Skin Roughness; Wrinkle; Fine Lines; Skin Thickness
Keywords: KB301; Wrinkles; Krystal Biotech; Décolletage; Lateral Canthal Lines; Décolleté; Pigmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KB301 (Active Comparator): non-integrating HSV-1 vector expressing human type III collagen
  Interventions: Biological: KB301
- Placebo (Placebo Comparator): sterile isotonic saline
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: KB301 — non-integrating HSV-1 vector expressing human type III collagen
  Arms: KB301
Other: Placebo — sterile isotonic saline
  Arms: Placebo

SUMMARY:
A Phase I Study of KB301, a Replication-Incompetent, Non-Integrating Vector Expressing Human Type III Collagen (COL3) for the Treatment of Superficial Skin Depressions

DETAILED DESCRIPTION:
Subjects enrolled in Cohort 1 will have a region of healthy buttock skin as a non-facial target area to receive two (2) injectable doses of KB301 (low or high). Cohort 1a will also present two regions of healthy buttock skin as a non-facial target area to receive two (2) injectable doses of KB301 (low or high) as well as a placebo injection. The objective of this cohort is to evaluate COL3A1 transgene expression (as measured by qRT-PCR of skin biopsies) and determine the optimal dose.

Subjects enrolled in Cohort 2 will present with bilaterally symmetrical regions of moderate to severe fine lines and skin roughness as the target areas; these areas will be randomly assigned to receive either KB301 or a placebo to determine the extent of skin improvement in the KB301 arm. Throughout the study subjects will complete questionnaires, have images captured of the target areas, undergo physical examinations, and have safety labs monitored.

Cohort 2 subjects may enroll in Cohort 2 extension, if they have not reverted back to baseline on the KB301 treated target area of the cheek. If subjects received KB301 to both cheek areas they will not be eligible for additional treatment and will be followed for durability. Subjects who received KB301 treatment to one cheek area, who have not reverted to baseline on the KB301 treated target area will be treated with KB301 on the cheek which previously received placebo. Subjects will be followed for durability, captured through investigator assessments, and questionnaires, while continuing to monitor safety.

Cohort 3 will be open label. Subjects will present with mild to moderate lateral canthal lines. The cohort will be split into two (3) subsets, Cohort 3a, Cohort 3b and Cohort 3c. Subjects in Cohort 3a and Cohort 3c will receive microinjections of KB301 and subjects in Cohort 3b will receive microneedling prior to topical application of KB301. Throughout the study, subjects will complete questionnaires, have images captured of the target areas, undergo physical examinations, and have assessment of improvement completed by the investigator. At Visit 5 the subject may begin retreatment with KB301 once weekly for three weeks and then will be followed for an additional 3 months, at the discretion of the investigator.

Cohort 4 will be open label. Subjects will present with dynamic décolleté wrinkles and/or pigmentation. Subjects in Cohort 4 will receive microinjections of KB301 to the décolleté area. Throughout the study, subjects will complete questionnaires, have images captured of the target areas, undergo physical examinations, and have assessment of improvement completed by the investigator. At Visit 5 the subject may begin retreatment with KB301 once weekly for three weeks and then will be followed for an additional 3 months, at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female in good general health, as determined by the investigator, aged ≥18 and ≤75 at the time of consent (only females for Cohort 4)
2. Regions of suitable skin to be selected as Target Area(s), as determined by a physical examination conducted by the investigator during the initial visit:

   * Cohort 1 - region of healthy buttock skin
   * Cohort 1a - bilaterally symmetric regions of healthy buttock skin at least 6 cm apart
   * Cohort 2 - bilaterally symmetric regions of moderate to severe fine lines and skin roughness (score of 2 or 3), as determined by investigator using the 5-point FLS and SRS on the cheeks above and below the zygomatic arch
   * Cohort 2 Extension- A subject who received a high dose regimen of KB301 to Target Areas below the zygomatic arch

     * Treatment group- Unilateral region of the cheek below the zygomatic arch, which was randomized to received placebo under Cohort 2, that per investigator assessment and consultation with the sponsor at Visit 1, is determined to be uneven as compared to the Target Area which received KB301
     * Observational group - Bilateral region of the cheeks below the zygomatic arch which were randomized to receive high dose 301 under Cohort 2 that show durability of KB301 to at least one of the two Target Areas
   * Cohort 3- Lateral canthal lines of mild to moderate severity at rest, per the Investigator's clinical assessment
   * Cohort 4- Dynamic décolleté wrinkles and /or pigmentation
3. A Fitzpatrick skin phototype score of I-IV
4. A negative pregnancy test at the Study Day 0 Visit for subjects of child-bearing potential and
5. Signed and dated informed consent and willingness to attend all study visits and complete all procedures required by this protocol.

Exclusion Criteria:

1. Any transient or chronic skin condition, disorder, or infection within 20 cm of the Target Areas at Day 0 that, in the opinion of the investigator, may confound study results
2. History of laser treatment or chemical peels to the Target Areas within six (6) months of the Study Day 0 Visit
3. History of surgical procedures to Target Areas, including removal of benign or malignant skin cancers that, in the opinion of the investigator, may confound study results
4. Administration of a cosmetic and/or clinical research investigational agent, at the location of the Target Areas within 6 months of the Study Day 0 Visit, that, in the opinion of the investigator, may confound study results
5. Scars, tattoos or tanned skin (defined as skin that is tanned from sun exposure or an applied skin color such as a spray tan) within the Target Area
6. Any condition (including a history or current evidence of substance abuse or dependence) that, in the investigator's opinion, would impact subject's ability to complete all study-related procedures and/or poses an additional risk to the assessment of safety of the Investigational Product
7. Women who are pregnant or nursing
8. Subject who is unwilling to comply with contraception requirements per-protocol
9. Subject is known to be noncompliant or is unlikely to comply with the requirements of the study protocol, in the opinion of the investigator.
10. Previously treated with KB301 under Cohorts 2, 2-extension, 3a, or 3b (Cohort 3c only)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of the safety profile of KB301 by recording adverse events using MedDRA System Organ Class and Preferred Term and collection of other clinical study procedures. | 4 months
  The primary outcome will look at the safety and tolerability of KB301 through the collection and quantification of adverse events, physical examinations, vital signs and clinical laboratory tests.

SECONDARY OUTCOMES:
Evaluation of COL3A1 transgene expression 2-days post-dose. | 12 months
  The secondary outcome measure in Cohorts 1 and 1a will compare a KB301 injection site biopsy, to an area of untreated healthy buttock skin biopsy (at least 6 cm away from the sites of KB301 injection), via qRT-PCR analysis.
Assessment of skin roughness as compared to baseline, using the Skin Roughness Scale (SRS). | 65 Days
  The secondary outcome measure in Cohort 2 will look at the mean change in the assessment of skin roughness as compared to baseline, using the Skin Roughness Scale (SRS). The SRS ranges from no fine lines (0) to extreme fine lines (4). A third-party independent blinded evaluator will perform the evaluations.
Assessment of fine line improvement as compared to baseline, using the Fine Lines Scale (FLS). | 65 Days
  The secondary outcome measure in Cohort 2, will look at the mean change in the assessment of fine lines as compared to baseline, using the Fine Lines Scale (FLS). The FLS ranges from no texture (0) to diffuse texture (4). A third-party independent blinded evaluator will perform the evaluations.
Subject assessment of aesthetic improvement over baseline, using the Subject Satisfaction Scale (SSS). | 65 Days
  The secondary outcome measure in Cohort 2, will look at the mean change in Subject's Satisfaction with the treatment per target area, as compared to baseline, using the Subject Satisfaction Scale (SSS), which is scored on a scale from 0-4, with 0 indicating not satisfied and 4 indicating excellent.
Assessment of skin fold thickness improvement over baseline, using a Caliper. | 65 Days
  The secondary outcome measure in Cohort 2, will look at the mean change in skinfold thickness of the non-facial target areas above the knee, using a Caliper to measure, as compared to baseline.
Subject assessment of aesthetic improvement over baseline, using the Subject Satisfaction Scale (SSS). | 3 Months
  The secondary outcome measure in Cohort 2 Extension, will look at the mean change in Subject's Satisfaction with the treatment per target area, as compared to baseline, using the Subject Satisfaction Scale (SSS), which is scored on a scale from 0-4, with 0 indicating not satisfied and 4 indicating excellent.
Investigator assessment of durability of high dose KB301, as compared to baseline. | 3 Months
  The secondary outcome measure in Cohort 2 Extension, will look at the durability of high dose KB301, as compared to baseline through an Investigator assessment.
Investigator assessment of global aesthetic improvement, as compared to baseline. | 4 Months
  The secondary outcome measure in Cohort 3 and Cohort 4 will look at the mean change in global aesthetic improvement, which is scored on a 5-point scale, ranging from much improved (2) to much worse (-2).
Subject assessment of global aesthetic improvement, as compared to baseline. | 4 Months
  The secondary outcome measure in Cohort 3 and Cohort 4 will look at the mean change in global aesthetic improvement, which is scored on a 5-point scale, ranging from much improved (2) to much worse (-2).
Subject treatment satisfaction as compared to baseline, using the Subject Satisfaction Questionnaire (SSQ). | 4 Months
  The secondary outcome measure in Cohort 3 and Cohort 4 will look at mean change in subject treatment satisfaction over baseline, using a 5-point Subject Satisfaction Questionnaire, ranging from very satisfied (2) to very dissatisfied (-2).

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Aesthetx, Campbell, California
  - Steve Yoelin, MD Medical Associates, Inc., Newport Beach, California
  - Mission Dermatology, Rancho Santa Margarita, California
  - Skin and Cancer Associates, LLP. D/B/A Center for Clinical and Cosmetic Research, Aventura, Florida

IPD SHARING:
Plan to Share IPD: No